CLINICAL TRIAL: NCT00600717
Title: Localizing Functional Brain Cortices and Epileptogenic Zones With High Frequency Brain Signals
Brief Title: Clinical Applications of High-Frequency Oscillations
Acronym: HFOs
Status: Withdrawn | Type: Observational
Why Stopped: No participants were enrolled to collected prospective data.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 2012-0866; 2018-8108; 2008-1439 (Other: CCHMC)
Record Dates: First submitted 2007-06-14; First posted 2008-01-25 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Epilepsy; Migraine; Headache; Pain; Autism; Cerebral Palsy; Brain Development; Traumatic Brain Injury; ADHD - Attention Deficit Disorder With Hyperactivity; Mental Health
Keywords: Magnetoencephalography(MEG); Electroencephalography (EEG); Intracranial recordings (iEEG/ECoG/SEEG); Functional Mapping; Epilepsy; Migraine; High frequency oscillations (HFOs); ripples; fast ripples; high-gamma; very high frequency oscillations (VHFOs); ultra fast oscillations; spikelet; fast spikelet; Optically Pumped Magnetometer; Wearable MEG; Multi-frequency Analysis; Frequency Encoded Source Imaging; Artificial Intelligence (AI); CUDA
MeSH Terms: conditions — Epilepsy; Migraine Disorders; Headache; Pain; Autistic Disorder; Cerebral Palsy; Brain Injuries, Traumatic; Attention Deficit Disorder with Hyperactivity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients and Healthy Children: Healthy children without dental works. Pediatric patients with epilepsy and migraine (headache).

SUMMARY:
The objective of this study is to utilize high-frequency brain signals (HFBS) to localize functional brain areas and characterize HFBS in epilepsy, migraine, and other brain disorders. Our goal is to create the world's first high-frequency MEG/EEG/ECoG/SEEG database for the developing brain. HFBS include high-gamma activation/oscillations, high-frequency oscillations (HFOs), ripples, fast ripples, spikelets, fast spikelets, and very high-frequency oscillations (VHFOs). While terminologies and frequency bands may vary among reports, both HFOs and high-gamma waves are crucial for understanding brain function and developing potential treatments for neurological disorders.

We have been developing an intelligent software platform to analyze signals from low to very high-frequency ranges across multiple frequency bands. To achieve these goals, we have developed several innovative techniques and software packages:

* Accumulated spectrogram
* Accumulated source imaging
* Frequency-encoded source imaging
* Multi-frequency analysis at source levels
* Artificial intelligence detection of HFOs
* Neural network analysis (Graph Theory)
* Other techniques (e.g., Independent Component Analysis, virtual sensors) These methods enable researchers to better understand the characteristics and significance of HFOs and high-gamma brain waves, contributing to advancements in the diagnosis and treatment of neurological disorders.

DETAILED DESCRIPTION:
The purpose of this study is to go beyond conventional analyses of brain signals in narrow frequency bands (typically 1-30 Hz) by measuring brain signals from infraslow to very fast frequencies (0.01 - 2800 Hz). Specifically, we propose to study physiological high-frequency oscillations (HFOs) in sensorimotor, auditory, visual, and language-evoked magnetic fields, and to investigate pathological HFOs in epilepsy, migraines, and other disorders. This is clinically important for several reasons.

For instance, there are 400,000 to 600,000 patients with refractory epilepsy in the United States. As these patients' seizures cannot be controlled by medication, epilepsy surgery is a potential cure. Accurate identification of ictogenic zones (the brain areas that cause seizures) is essential for favorable surgical outcomes. Unfortunately, the existing method, electrocorticography (ECoG), requires placing electrodes on the brain surface to capture spikes (typically, 14-70 Hz), which is both risky and costly. Our study aims to use magnetoencephalography (MEG) and electroencephalography (EEG) to identify ictogenic zones non-invasively. To achieve this goal, we propose detecting high-frequency (70-2500 Hz) and low-frequency (< 14 Hz) brain signals using advanced signal processing methods. Our central hypothesis is that high-frequency brain signals will lead to significantly improved rates of seizure freedom compared to spikes. This hypothesis is based on recent reports that high-frequency brain signals are localized to ictogenic zones.

Leveraging our unique resources and expertise, we plan to address four specific aims:

1. Quantify the Spatial Concordance: We will quantify the spatial concordance between MEG and ECoG signals in both low and high-frequency ranges. We hypothesize that ictogenic zones determined by invasive ECoG can be non-invasively detected and localized by high-frequency MEG signals.
2. Quantify the Occurrence Concordance: We will quantify the occurrence concordance between EEG and ECoG signals in both low and high-frequency ranges. We hypothesize that epileptic high-frequency signals from the ictogenic zones determined by invasive ECoG can also be non-invasively detected by EEG, although the localization of EEG may be significantly inferior to that of MEG.
3. Improve Epilepsy Surgery Outcomes: We will determine whether epilepsy surgery based on multi-frequency signals (low-frequency brain signals, spikes, and high-frequency brain signals), instead of spikes alone, leads to better seizure outcomes. We hypothesize that epilepsy surgery guided by high-frequency brain signals detected with MEG/EEG will significantly improve surgical outcomes.
4. Enhance Pre-surgical Planning: We will determine whether multi-frequency analyses provide more information than single-frequency analysis for estimating epileptogenic zones for pre-surgical ECoG electrode implantation. We hypothesize that covering all brain areas generating low to high-frequency epileptic activity is a prerequisite to localize multiple ictogenic zones for favorable post-surgical outcomes.

To yield definitive results, we propose a multi-center study to determine if high-frequency brain signals are new biomarkers for significantly improving epilepsy surgery outcomes. According to our pilot data, localization of epileptogenic zones with MEG high-frequency signals can increase post-operative seizure freedom by approximately 30-40%. The proposed study should result in millions of intractable epilepsy patients being seizure-free. Additionally, this study lays the foundation for using low and high-frequency brain signals as new biomarkers for the diagnosis and treatment of various other disorders (e.g., migraine, autism).

Furthermore, we will incorporate Optically Pumped Magnetometers MEG (OPM-MEG) to enhance the detection of high-frequency brain signals. OPM-MEG offers higher sensitivity and spatial resolution compared to conventional MEG, making it an invaluable tool for our research objectives.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and cooperative.
* Ages: from 1 day to 69 years (male or female).
* Normal hearing and vision.
* Normal hand movement.
* No history of neurological or psychiatric diseases.
* No family history of genetic neurological or psychiatric diseases.
* No metal implants such as pacemakers, neuro-stimulators, cochlear implants, etc.

Exclusion Criteria:

* Taking any medications for depression, neurologic, or psychiatric conditions.
* Not feeling well, having epilepsy, or other brain disorders.
* Recent concussion or head injury.
* Presence of metal in the body, such as dental braces, which could cause "magnetic noise". A simple, quick "magnetic noise screening" can be conducted at the MEG Center to determine eligibility.
* Presence of electrical or metal implants such as pacemakers, neuro-stimulators, or orthopedic pins or plates. The research nurse will discuss all exclusions in further detail before the magnetic resonance imaging (MRI) scan.
* Inability to pass the pre-experimental screening.

Ages: 1 Day to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will obtain MEG/EEG data from healthy subjects, recruiting only individuals without underlying health conditions. Additionally, this study will utilize clinical MEG/EEG data from patients, which are acquired as part of standard clinical care for clinical purposes. Since women, girls, and minorities are included in the population to whom recruiting materials are directed, we anticipate that subject selection will be equitable.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2000-11-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
epileptic foci | one year
  Accuracy of localization of epileptic foci

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xiang, Ph.D M.D., Study Director — Children's Hospital Medical Center, Cincinnati
Locations (1):
- MEG, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kotecha R, Xiang J, Wang Y, Huo X, Hemasilpin N, Fujiwara H, Rose D, deGrauw T. Time, frequency and volumetric differences of high-frequency neuromagnetic oscillation between left and right somatosensory cortices. Int J Psychophysiol. 2009 May;72(2):102-10. doi: 10.1016/j.ijpsycho.2008.10.009. Epub 2008 Nov 14. PMID 19041674
- [Background] Wang Y, Xiang J, Kotecha R, Vannest J, Liu Y, Rose D, Schapiro M, Degrauw T. Spatial and frequency differences of neuromagnetic activities between the perception of open- and closed-class words. Brain Topogr. 2008 Dec;21(2):75-85. doi: 10.1007/s10548-008-0060-7. Epub 2008 Aug 5. PMID 18679788
- [Background] Liu Y, Xiang J, Wang Y, Vannest JJ, Byars AW, Rose DF. Spatial and frequency differences of neuromagnetic activities in processing concrete and abstract words. Brain Topogr. 2008 Spring;20(3):123-9. doi: 10.1007/s10548-007-0038-x. Epub 2007 Dec 6. PMID 18058218
- [Background] Xiang J, Xiao Z. Spatiotemporal and frequency signatures of noun and verb processing: a wavelet-based beamformer study. J Clin Exp Neuropsychol. 2009 Aug;31(6):648-57. doi: 10.1080/13803390802448651. Epub 2008 Dec 22. PMID 19105073
- [Background] Guo X, Xiang J, Mun-Bryce S, Bryce M, Huang S, Huo X, Wang Y, Rose D, Degrauw T, Gartner K, Song T, Schmit J, Vargus-Adams J. Aberrant high-gamma oscillations in the somatosensory cortex of children with cerebral palsy: a meg study. Brain Dev. 2012 Aug;34(7):576-83. doi: 10.1016/j.braindev.2011.09.012. Epub 2011 Oct 21. PMID 22018901
- [Background] Korostenskaja M, Pardos M, Kujala T, Rose DF, Brown D, Horn P, Wang Y, Fujiwara H, Xiang J, Kabbouche MA, Powers SW, Hershey AD. Impaired auditory information processing during acute migraine: a magnetoencephalography study. Int J Neurosci. 2011 Jul;121(7):355-65. doi: 10.3109/00207454.2011.560312. Epub 2011 Mar 22. PMID 21425948
- [Background] Zhang R, Wu T, Wang Y, Liu H, Zou Y, Liu W, Xiang J, Xiao C, Yang L, Fu Z. Interictal magnetoencephalographic findings related with surgical outcomes in lesional and nonlesional neocortical epilepsy. Seizure. 2011 Nov;20(9):692-700. doi: 10.1016/j.seizure.2011.06.021. Epub 2011 Jul 22. PMID 21782477
- [Background] Wang Y, Xiang J, Vannest J, Holroyd T, Narmoneva D, Horn P, Liu Y, Rose D, deGrauw T, Holland S. Neuromagnetic measures of word processing in bilinguals and monolinguals. Clin Neurophysiol. 2011 Sep;122(9):1706-17. doi: 10.1016/j.clinph.2011.02.008. Epub 2011 Mar 16. PMID 21414839
- [Background] Korostenskaja M, Pardos M, Fujiwara H, Kujala T, Horn P, Rose D, Byars A, Brown D, Seo JH, Wang Y, Vannest J, Xiang J, Degrauw T, Naatanen R, Lee KH. Neuromagnetic evidence of impaired cortical auditory processing in pediatric intractable epilepsy. Epilepsy Res. 2010 Nov;92(1):63-73. doi: 10.1016/j.eplepsyres.2010.08.008. Epub 2010 Sep 21. PMID 20863661
- [Background] Meng L, Xiang J, Kotecha R, Rose D, Zhao H, Zhao D, Yang J, Degrauw T. White matter abnormalities in children and adolescents with temporal lobe epilepsy. Magn Reson Imaging. 2010 Nov;28(9):1290-8. doi: 10.1016/j.mri.2010.03.046. Epub 2010 Jul 24. PMID 20656430
- [Background] Huo X, Wang Y, Kotecha R, Kirtman EG, Fujiwara H, Hemasilpin N, Degrauw T, Rose DF, Xiang J. High gamma oscillations of sensorimotor cortex during unilateral movement in the developing brain: a MEG study. Brain Topogr. 2011 Jan;23(4):375-84. doi: 10.1007/s10548-010-0151-0. Epub 2010 Jun 25. PMID 20577795
- [Background] Wang X, Xiang J, Wang Y, Pardos M, Meng L, Huo X, Korostenskaja M, Powers SW, Kabbouche MA, Hershey AD. Identification of abnormal neuromagnetic signatures in the motor cortex of adolescent migraine. Headache. 2010 Jun;50(6):1005-16. doi: 10.1111/j.1526-4610.2010.01674.x. Epub 2010 May 7. PMID 20487034
- [Background] Chen Y, Xiang J, Kirtman EG, Wang Y, Kotecha R, Liu Y. Neuromagnetic biomarkers of visuocortical development in healthy children. Clin Neurophysiol. 2010 Sep;121(9):1555-1562. doi: 10.1016/j.clinph.2010.03.029. Epub 2010 Apr 14. PMID 20395171
- [Background] Huo X, Xiang J, Wang Y, Kirtman EG, Kotecha R, Fujiwara H, Hemasilpin N, Rose DF, Degrauw T. Gamma oscillations in the primary motor cortex studied with MEG. Brain Dev. 2010 Sep;32(8):619-24. doi: 10.1016/j.braindev.2009.09.021. PMID 19836911
- [Background] Xiang J, Liu Y, Wang Y, Kirtman EG, Kotecha R, Chen Y, Huo X, Fujiwara H, Hemasilpin N, Lee K, Mangano FT, Leach J, Jones B, DeGrauw T, Rose D. Frequency and spatial characteristics of high-frequency neuromagnetic signals in childhood epilepsy. Epileptic Disord. 2009 Jun;11(2):113-25. doi: 10.1684/epd.2009.0253. Epub 2009 May 27. PMID 19473946
- [Background] Xiang J, Liu Y, Wang Y, Kotecha R, Kirtman EG, Chen Y, Huo X, Fujiwara H, Hemasilpin N, DeGrauw T, Rose D. Neuromagnetic correlates of developmental changes in endogenous high-frequency brain oscillations in children: a wavelet-based beamformer study. Brain Res. 2009 Jun 5;1274:28-39. doi: 10.1016/j.brainres.2009.03.068. Epub 2009 Apr 9. PMID 19362072
- [Background] Leiken KA, Xiang J, Curry E, Fujiwara H, Rose DF, Allen JR, Kacperski JE, O'Brien HL, Kabbouche MA, Powers SW, Hershey AD. Quantitative neuromagnetic signatures of aberrant cortical excitability in pediatric chronic migraine. J Headache Pain. 2016;17:46. doi: 10.1186/s10194-016-0641-x. Epub 2016 Apr 26. PMID 27113076
- [Background] Meng L, Xiang J. Frequency specific patterns of resting-state networks development from childhood to adolescence: A magnetoencephalography study. Brain Dev. 2016 Nov;38(10):893-902. doi: 10.1016/j.braindev.2016.05.004. Epub 2016 Jun 7. PMID 27287665
- [Background] Li F, Xiang J, Wu T, Zhu D, Shi J. Abnormal resting-state brain activity in headache-free migraine patients: A magnetoencephalography study. Clin Neurophysiol. 2016 Aug;127(8):2855-2861. doi: 10.1016/j.clinph.2016.05.015. Epub 2016 May 26. PMID 27417062
- [Background] Wu D, Zhou Y, Xiang J, Tang L, Liu H, Huang S, Wu T, Chen Q, Wang X. Multi-frequency analysis of brain connectivity networks in migraineurs: a magnetoencephalography study. J Headache Pain. 2016;17:38. doi: 10.1186/s10194-016-0636-7. Epub 2016 Apr 18. PMID 27090418
- [Background] Xiang J, Leiken K, Degrauw X, Kay B, Fujiwara H, Rose DF, Allen JR, Kacperski JE, O'Brien HL, Kabbouche MA, Powers SW, Hershey AD. Spatial Heterogeneity of Cortical Excitability in Migraine Revealed by Multifrequency Neuromagnetic Signals. J Pain. 2016 Jun;17(6):694-706. doi: 10.1016/j.jpain.2016.02.009. Epub 2016 Mar 10. PMID 26970516
- [Background] Tang L, Xiang J, Huang S, Miao A, Ge H, Liu H, Wu D, Guan Q, Wu T, Chen Q, Yang L, Lu X, Hu Z, Wang X. Neuromagnetic high-frequency oscillations correlate with seizure severity in absence epilepsy. Clin Neurophysiol. 2016 Feb;127(2):1120-1129. doi: 10.1016/j.clinph.2015.08.016. Epub 2015 Sep 5. PMID 26384756
- [Background] Pardos M, Korostenskaja M, Xiang J, Fujiwara H, Lee KH, Horn PS, Byars A, Vannest J, Wang Y, Hemasilpin N, Rose DF. Physical Feature Encoding and Word Recognition Abilities Are Altered in Children with Intractable Epilepsy: Preliminary Neuromagnetic Evidence. Behav Neurol. 2015;2015:237436. doi: 10.1155/2015/237436. Epub 2015 Jun 3. PMID 26146459
- [Background] Liu H, Ge H, Xiang J, Miao A, Tang L, Wu T, Chen Q, Yang L, Wang X. Resting state brain activity in patients with migraine: a magnetoencephalography study. J Headache Pain. 2015;16:525. doi: 10.1186/s10194-015-0525-5. Epub 2015 May 7. PMID 25968099
- [Background] Xiang J, Korostenskaja M, Molloy C, deGrauw X, Leiken K, Gilman C, Meinzen-Derr J, Fujiwara H, Rose DF, Mitchell T, Murray DS. Multi-frequency localization of aberrant brain activity in autism spectrum disorder. Brain Dev. 2016 Jan;38(1):82-90. doi: 10.1016/j.braindev.2015.04.007. Epub 2015 Apr 27. PMID 25937458
- [Background] Leiken K, Xiang J, Zhang F, Shi J, Tang L, Liu H, Wang X. Magnetoencephalography detection of high-frequency oscillations in the developing brain. Front Hum Neurosci. 2014 Dec 12;8:969. doi: 10.3389/fnhum.2014.00969. eCollection 2014. PMID 25566015
- [Background] Xiang J, Korman A, Samarasinghe KM, Wang X, Zhang F, Qiao H, Sun B, Wang F, Fan HH, Thompson EA. Volumetric imaging of brain activity with spatial-frequency decoding of neuromagnetic signals. J Neurosci Methods. 2015 Jan 15;239:114-28. doi: 10.1016/j.jneumeth.2014.10.007. Epub 2014 Oct 18. PMID 25455340
- [Background] Xiang J, Tenney JR, Korman AM, Leiken K, Rose DF, Harris E, Yuan W, Horn PS, Holland K, Loring DW, Glauser TA. Quantification of Interictal Neuromagnetic Activity in Absence Epilepsy with Accumulated Source Imaging. Brain Topogr. 2015 Nov;28(6):904-14. doi: 10.1007/s10548-014-0411-5. Epub 2014 Oct 31. PMID 25359158
- [Background] Tenney JR, Fujiwara H, Horn PS, Vannest J, Xiang J, Glauser TA, Rose DF. Low- and high-frequency oscillations reveal distinct absence seizure networks. Ann Neurol. 2014 Oct;76(4):558-67. doi: 10.1002/ana.24231. Epub 2014 Sep 8. PMID 25042348
- [Background] Xiang J, Luo Q, Kotecha R, Korman A, Zhang F, Luo H, Fujiwara H, Hemasilpin N, Rose DF. Accumulated source imaging of brain activity with both low and high-frequency neuromagnetic signals. Front Neuroinform. 2014 May 21;8:57. doi: 10.3389/fninf.2014.00057. eCollection 2014. PMID 24904402
- [Background] Ge HT, Liu HX, Xiang J, Miao AL, Tang L, Guan QS, Wu T, Chen QQ, Yang L, Wang XS. Abnormal cortical activation in females with acute migraine: a magnetoencephalography study. Clin Neurophysiol. 2015 Jan;126(1):170-9. doi: 10.1016/j.clinph.2014.03.033. Epub 2014 Apr 16. PMID 24854723
- [Background] Miao A, Xiang J, Tang L, Ge H, Liu H, Wu T, Chen Q, Hu Z, Lu X, Wang X. Using ictal high-frequency oscillations (80-500Hz) to localize seizure onset zones in childhood absence epilepsy: a MEG study. Neurosci Lett. 2014 Apr 30;566:21-6. doi: 10.1016/j.neulet.2014.02.038. Epub 2014 Feb 26. PMID 24582907
- [Background] Miao A, Tang L, Xiang J, Guan Q, Ge H, Liu H, Wu T, Chen Q, Yang L, Lu X, Hu Z, Wang X. Dynamic magnetic source imaging of absence seizure initialization and propagation: a magnetoencephalography study. Epilepsy Res. 2014 Mar;108(3):468-80. doi: 10.1016/j.eplepsyres.2014.01.006. Epub 2014 Jan 29. PMID 24534760
- [Background] Xiang J, Degrauw X, Korman AM, Allen JR, O'Brien HL, Kabbouche MA, Powers SW, Hershey AD. Neuromagnetic abnormality of motor cortical activation and phases of headache attacks in childhood migraine. PLoS One. 2013 Dec 27;8(12):e83669. doi: 10.1371/journal.pone.0083669. eCollection 2013. PMID 24386250
- [Background] Xiang J, deGrauw X, Korostenskaja M, Korman AM, O'Brien HL, Kabbouche MA, Powers SW, Hershey AD. Altered cortical activation in adolescents with acute migraine: a magnetoencephalography study. J Pain. 2013 Dec;14(12):1553-63. doi: 10.1016/j.jpain.2013.04.009. Epub 2013 Jun 21. PMID 23792072
- [Background] Korostenskaja M, Harris E, Giovanetti C, Horn P, Wang Y, Rose D, Fujiwara H, Xiang J. Magnetoencephalography reveals altered auditory information processing in youth with obsessive-compulsive disorder. Psychiatry Res. 2013 May 30;212(2):132-40. doi: 10.1016/j.pscychresns.2012.11.011. Epub 2013 Mar 30. PMID 23545237
- [Background] Song PP, Xiang J, Jiang L, Chen HS, Liu BK, Hu Y. Dynamic Changes in Spectral and Spatial Signatures of High Frequency Oscillations in Rat Hippocampi during Epileptogenesis in Acute and Chronic Stages. Front Neurol. 2016 Nov 28;7:204. doi: 10.3389/fneur.2016.00204. eCollection 2016. PMID 27965619
- [Background] Wu C, Xiang J, Sun J, Huang S, Tang L, Miao A, Zhou Y, Chen Q, Hu Z, Wang X. Quantify neuromagnetic network changes from pre-ictal to ictal activities in absence seizures. Neuroscience. 2017 Aug 15;357:134-144. doi: 10.1016/j.neuroscience.2017.05.038. Epub 2017 May 31. PMID 28576731
- [Background] Wu C, Xiang J, Jiang W, Huang S, Gao Y, Tang L, Zhou Y, Wu D, Chen Q, Hu Z, Wang X. Altered Effective Connectivity Network in Childhood Absence Epilepsy: A Multi-frequency MEG Study. Brain Topogr. 2017 Sep;30(5):673-684. doi: 10.1007/s10548-017-0555-1. Epub 2017 Mar 12. PMID 28286918
- [Background] Chen D, Wan S, Xiang J, Bao FS. A high-performance seizure detection algorithm based on Discrete Wavelet Transform (DWT) and EEG. PLoS One. 2017 Mar 9;12(3):e0173138. doi: 10.1371/journal.pone.0173138. eCollection 2017. PMID 28278203
- [Background] Feng YG; Xiang J; Wu J; Zhu D. Clinical application of magnetoencephalography with high frequency oscillations in epilepsy. Chin J Neuromed.2017; 16(10): 973-977
- [Background] Du, J ; Shan, Y ; Li, L ; Fan, X ; An, Y ; Zhang, X; Xiang, ; Ren, L ; Wang, Y. Dynamic Propagation of Interictal Epileptic Spike of Medial Temporal Lobe Epilepsy Predict Seizure Network: A MEG combined with SEEG Study. Epilepsia, 2017, 58(SI, 5): 871
- [Background] Wu J, Feng YG; Liu PF, Tan JL, Yan XQ, Zhu D, Xiang J. High frequency magnetoencephalographic signals in surgery of refractory temporal lobe epilepsy. Chin J Neuromed, 2017, 16(6): 620-624
- [Background] Fan Y, Xiang J, Yang K. Multi-frequency analysis of neuromagnetic activity between eyes-open and eyes-closed in the developing brain. The Journal of Japan Biomagnetism and Bioelectromagnetics Society. 2017 May 20; 30(1):90
- [Background] Wang F, wang XW, Yu T, Xiang J, Hu Y. Multi-band frequency analysis of neuromagnetic signals from primary epileptogenic foci and mirror foci. The Journal of Japan Biomagnetism and Bioelectromagnetics Society. 2017 May 20; 30(1):64.
- [Background] Liang C, Earl B, Thompson I, Whitaker K, Cahn S, Xiang J, Fu QJ, Zhang F. Musicians Are Better than Non-musicians in Frequency Change Detection: Behavioral and Electrophysiological Evidence. Front Neurosci. 2016 Oct 25;10:464. doi: 10.3389/fnins.2016.00464. eCollection 2016. PMID 27826221
- [Background] Qiu W, Yu C, Gao Y, Miao A, Tang L, Huang S, Jiang W, Sun J, Xiang J, Wang X. Disrupted topological organization of structural brain networks in childhood absence epilepsy. Sci Rep. 2017 Sep 20;7(1):11973. doi: 10.1038/s41598-017-10778-0. PMID 28931825
- [Background] Al-Marri F, Reza F, Begum T, Hitam WHW, Jin GK, Xiang J. Neural activation patterns and connectivity in visual attention during Number and Non-number processing: An ERP study using the Ishihara pseudoisochromatic plates. J Integr Neurosci. 2017 Oct 25. doi: 10.3233/JIN-170058. Online ahead of print. PMID 29081422
- [Background] Wu T, Zhang L, Wan S, Chen D, Xiang J, Shi Y, Chen Q, Zhang R, Jiang T, Liu H. Magnetoencephalography (MEG): A noninvasive technique for surgical treatment of epilepsy. Science. 2017 December 27; 358(6370):25
- [Background] Xiang J, Leiken K, Assessment of epileptogenicity of multi-frequency neuromagnetic activity with frequency-encoded magnetic source imaging. The Journal of Japan Biomagnetism and Bioelectromagnetics Society. 2017 May 20; 30(1):39
- [Background] Dinga S, Wu D, Huang S, Wu C, Wang X, Shi J, Hu Y, Liang C, Zhang F, Lu M, Leiken K, Xiang J. Neuromagnetic correlates of audiovisual word processing in the developing brain. Int J Psychophysiol. 2018 Jun;128:7-21. doi: 10.1016/j.ijpsycho.2018.03.016. Epub 2018 Mar 23. PMID 29580903
- [Background] Tenney JR, Kadis DS, Agler W, Rozhkov L, Altaye M, Xiang J, Vannest J, Glauser TA. Ictal connectivity in childhood absence epilepsy: Associations with outcome. Epilepsia. 2018 May;59(5):971-981. doi: 10.1111/epi.14067. Epub 2018 Apr 6. PMID 29633248
- [Background] Guo J, Yang K, Liu H, Yin C, Xiang J, Li H, Ji R, Gao Y. A Stacked Sparse Autoencoder-Based Detector for Automatic Identification of Neuromagnetic High Frequency Oscillations in Epilepsy. IEEE Trans Med Imaging. 2018 Nov;37(11):2474-2482. doi: 10.1109/TMI.2018.2836965. Epub 2018 May 15. PMID 29994761
- [Background] Ishii R, Pascual-Marqui RD, Canuet L, Xiang J, Gaetz WC. Editorial: New Insights on Basic and Clinical Aspects of EEG and MEG Connectome. Front Hum Neurosci. 2018 Jun 5;12:232. doi: 10.3389/fnhum.2018.00232. eCollection 2018. No abstract available. PMID 29922140
- [Background] Ran X, Xiang J, Song PP, Jiang L, Liu BK, Hu Y. Effects of gap junctions blockers on fast ripples and connexin in rat hippocampi after status epilepticus. Epilepsy Res. 2018 Oct;146:28-35. doi: 10.1016/j.eplepsyres.2018.07.010. Epub 2018 Jul 20. PMID 30056318
- [Background] Wu T, Fan J, Chen Y, Xiang J, Zhu D, Zhang J, Shi J, Jiang T. Interictal Abnormalities of Neuromagnetic Gamma Oscillations in Migraine Following Negative Emotional Stimulation. Front Behav Neurosci. 2018 Aug 17;12:169. doi: 10.3389/fnbeh.2018.00169. eCollection 2018. PMID 30174594
- [Background] Miao A, Wang Y, Xiang J, Liu Q, Chen Q, Qiu W, Liu H, Tang L, Gao Y, Wu C, Yu Y, Sun J, Jiang W, Shi Q, Zhang T, Hu Z, Wang X. Ictal Source Locations and Cortico-Thalamic Connectivity in Childhood Absence Epilepsy: Associations with Treatment Response. Brain Topogr. 2019 Jan;32(1):178-191. doi: 10.1007/s10548-018-0680-5. Epub 2018 Oct 5. PMID 30291582
- [Background] Zhou ZY, Yu YW, Wu D, Liu HX, Xiang J, Wu T, Chen QQ, Wang XS. Abnormality of visual neuromagnetic activation in female migraineurs without aura between attacks. J Headache Pain. 2019 Jan 16;20(1):7. doi: 10.1186/s10194-018-0957-9. PMID 30651072
- [Background] Ren J, Xiang J, Chen Y, Li F, Wu T, Shi J. Abnormal functional connectivity under somatosensory stimulation in migraine: a multi-frequency magnetoencephalography study. J Headache Pain. 2019 Jan 9;20(1):3. doi: 10.1186/s10194-019-0958-3. PMID 30626318
- [Background] Yang K, Chen J, Xiang J, Liu H, Zou Y, Kan W, Liu Y, Li L. Histopathologic and Clinical Correlation of Aberrant Neuromagnetic Activities with Low to High Frequency of Gliomas. World Neurosurg. 2019 Mar;123:e609-e620. doi: 10.1016/j.wneu.2018.11.235. Epub 2018 Dec 8. PMID 30529596
- [Background] Meng L, Xiang J. Brain Network Analysis and Classification Based on Convolutional Neural Network. Front Comput Neurosci. 2018 Dec 10;12:95. doi: 10.3389/fncom.2018.00095. eCollection 2018. PMID 30618690
- [Background] Leng X, Xiang J, Yang Y, Yu T, Qi X, Zhang X, Wu S, Wang Y. Frequency-specific changes in the default mode network in patients with cingulate gyrus epilepsy. Hum Brain Mapp. 2020 Jun 15;41(9):2447-2459. doi: 10.1002/hbm.24956. Epub 2020 Feb 25. PMID 32096905
- [Background] Shi Q, Zhang T, Miao A, Sun J, Sun Y, Chen Q, Hu Z, Xiang J, Wang X. Differences Between Interictal and Ictal Generalized Spike-Wave Discharges in Childhood Absence Epilepsy: A MEG Study. Front Neurol. 2020 Jan 24;10:1359. doi: 10.3389/fneur.2019.01359. eCollection 2019. PMID 32038453
- [Background] Yin C, Zhang X, Xiang J, Chen Z, Li X, Wu S, Lv P, Wang Y. Altered effective connectivity network in patients with insular epilepsy: A high-frequency oscillations magnetoencephalography study. Clin Neurophysiol. 2020 Feb;131(2):377-384. doi: 10.1016/j.clinph.2019.11.021. Epub 2019 Dec 6. PMID 31865139
- [Background] Jiang W, Wu C, Xiang J, Miao A, Qiu W, Tang L, Huang S, Chen Q, Hu Z, Wang X. Dynamic Neuromagnetic Network Changes of Seizure Termination in Absence Epilepsy: A Magnetoencephalography Study. Front Neurol. 2019 Jul 2;10:703. doi: 10.3389/fneur.2019.00703. eCollection 2019. PMID 31338058
- [Background] Liang C, Wenstrup LH, Samy RN, Xiang J, Zhang F. The Effect of Side of Implantation on the Cortical Processing of Frequency Changes in Adult Cochlear Implant Users. Front Neurosci. 2020 Apr 29;14:368. doi: 10.3389/fnins.2020.00368. eCollection 2020. PMID 32410947
- [Background] Firestone GM, McGuire K, Liang C, Zhang N, Blankenship CM, Xiang J, Zhang F. A Preliminary Study of the Effects of Attentive Music Listening on Cochlear Implant Users' Speech Perception, Quality of Life, and Behavioral and Objective Measures of Frequency Change Detection. Front Hum Neurosci. 2020 Mar 31;14:110. doi: 10.3389/fnhum.2020.00110. eCollection 2020. PMID 32296318
- [Background] Xiang J, Maue E, Fan Y, Qi L, Mangano FT, Greiner H, Tenney J. Kurtosis and skewness of high-frequency brain signals are altered in paediatric epilepsy. Brain Commun. 2020 Mar 31;2(1):fcaa036. doi: 10.1093/braincomms/fcaa036. eCollection 2020. PMID 32954294
- [Background] Xiang J, Maue E, Tong H, Mangano FT, Greiner H, Tenney J. Neuromagnetic high frequency spikes are a new and noninvasive biomarker for localization of epileptogenic zones. Seizure. 2021 Jul;89:30-37. doi: 10.1016/j.seizure.2021.04.024. Epub 2021 May 4. PMID 33975080
- [Background] Xiang J, Maue E, Fujiwara H, Mangano FT, Greiner H, Tenney J. Delineation of epileptogenic zones with high frequency magnetic source imaging based on kurtosis and skewness. Epilepsy Res. 2021 May;172:106602. doi: 10.1016/j.eplepsyres.2021.106602. Epub 2021 Mar 8. PMID 33713889
- [Background] Xiang J, Yu X, Bonnette S, Anand M, Riehm CD, Schlink B, Diekfuss JA, Myer GD, Jiang Y. Improved Biomagnetic Signal-To-Noise Ratio and Source Localization Using Optically Pumped Magnetometers with Synthetic Gradiometers. Brain Sci. 2023 Apr 15;13(4):663. doi: 10.3390/brainsci13040663. PMID 37190628
- [Background] Xiang J, Tong H, Jiang Y, Barnes-Davis ME. Spatial and Frequency Specific Artifact Reduction in Optically Pumped Magnetometer Recordings. J Integr Neurosci. 2022 Aug 16;21(5):145. doi: 10.31083/j.jin2105145. PMID 36137963
- [Background] Chen D, Liu K, Guo J, Bi L, Xiang J. Editorial: Brain-computer interface and its applications. Front Neurorobot. 2023 Feb 9;17:1140508. doi: 10.3389/fnbot.2023.1140508. eCollection 2023. No abstract available. PMID 36845071
- [Background] Zhang F, Han JH, Samy R, Xiang J. Editorial: Changes in the auditory brain following deafness, cochlear implantation, and auditory training, volume II. Front Hum Neurosci. 2023 Feb 6;17:1124304. doi: 10.3389/fnhum.2023.1124304. eCollection 2023. No abstract available. PMID 36814434
- [Background] Guo J, Xiao N, Li H, He L, Li Q, Wu T, He X, Chen P, Chen D, Xiang J, Peng X. Transformer-Based High-Frequency Oscillation Signal Detection on Magnetoencephalography From Epileptic Patients. Front Mol Biosci. 2022 Mar 4;9:822810. doi: 10.3389/fmolb.2022.822810. eCollection 2022. PMID 35309504
- [Background] Sun Y, Li Y, Sun J, Zhang K, Tang L, Wu C, Gao Y, Liu H, Huang S, Hu Z, Xiang J, Wang X. Functional reorganization of brain regions into a network in childhood absence epilepsy: A magnetoencephalography study. Epilepsy Behav. 2021 Sep;122:108117. doi: 10.1016/j.yebeh.2021.108117. Epub 2021 Jul 8. PMID 34246893
- [Background] Sun K, Yu T, Yang D, Ren Z, Qiao L, Ni D, Wang X, Zhao Y, Chen X, Xiang J, Chen N, Gao R, Yang K, Lin Y, Kober T, Zhang G. Fluid and White Matter Suppression Imaging and Voxel-Based Morphometric Analysis in Conventional Magnetic Resonance Imaging-Negative Epilepsy. Front Neurol. 2021 Apr 29;12:651592. doi: 10.3389/fneur.2021.651592. eCollection 2021. PMID 33995250
- [Result] Xiang J, Ishii R, Yang X. Editorial: High Frequency Brain Signals: From Basic Research to Clinical Application. Front Hum Neurosci. 2022 Mar 30;16:872478. doi: 10.3389/fnhum.2022.872478. eCollection 2022. No abstract available. PMID 35431837
- See also: Xiang Lab's website offers in-depth insights into both basic scientific research and its clinical applications. — http://www.cincinnatichildrens.org/research/div/neurology/labs/xiang-lab/
- See also: The GitHub website offers extensive resources on software, methodologies, manuals, guides, and other information for analyzing signals across various frequency bands, ranging from low to high. — https://github.com/brainx888